CLINICAL TRIAL: NCT07301021
Title: Velopharyngeal Insufficiency After Maxillomandibular Advancement Osteotomy in Obstructive Sleep Apnea Patients
Acronym: VPIMMA
Status: Not yet recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. J. de Lange, MD DMD, Prof.dr. Jan de Lange, Head of Department Oral and Maxillofacial Surgery (Amsterdam UMC), Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL83076.018.23
Record Dates: First submitted 2025-07-30; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Velopharyngeal Insufficiency; Swallowing; Nasality; Speech
Keywords: maxillomandibular advancement; obstructive sleep apnea; velopharyngeal insufficiency; speech therapy; swallowing; nasality; speech
MeSH Terms: conditions — Velopharyngeal Insufficiency; Speech; Sleep Apnea, Obstructive; Communication Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSA patients after an MMA: Patients with obstructive sleep apnea (OSA) who underwent a maxillomandibular advancement (MMA)

SUMMARY:
The aim of this study is to gain insight into the development of velopharyngeal insufficiency (VPI) in patients who have undergone maxillomandibular advancement osteotomy (MMA) as a treatment for obstructive sleep apnea syndrome (OSAS). A speech therapist evaluates nasality, speech, and swallowing before and after the surgery.

DETAILED DESCRIPTION:
This study will be conducted at Amsterdam UMC. Adult patients with mild to severe obstructive sleep apnea syndrome (OSAS) who are eligible for maxillomandibular advancement (MMA) surgery will be invited to participate in this prospective cohort study. Patients will be evaluated by two speech therapists at four different time points: before surgery (T0), 6 weeks after surgery (T1), 3 months after surgery (T2), 6 months after surgery (T3) and 1 year after surgery (T4).

Patients will undergo objective assessments focusing on three components: nasality, speech, and swallowing. The Nasometer, a non-invasive analysis tool, will be used to measure the presence of nasality in speech production. Speech will be scored using the Cleft Audit Protocol for Speech - Augmented (CAPS-A), an instrument where speech therapists evaluate various aspects of speech performance. Swallowing will be assessed using the Functional Oral Intake Scale (FOIS), a scoring system that evaluates patients' swallowing abilities. Additionally, the swallowing speed/volume test will measure how quickly and how much water a patient can swallow. Thereby, for the subjective evaluation patients will receive the following questionnaires by email: OHIP-14 (oral health related quality of life), FOSQ (functional outcomes of sleep questionnaire), and the NSD (neurosensory disturbance questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Mild to severe OSA
* Indication for MMA for OSA treatment

Exclusion Criteria:

* patients who underwent other adjunctive procedures at the time of MMA (e.g., multipiece le Fort osteotomy, TMJ reconstruction
* Previous history of orthognathic surgery
* Previous history of orthognathic surgery
* Previous history of oropharyngeal surgery (UPPP or multi-level surgery)
* Cleft palate and syndromic patients
* Neuromusculair diseases which causes VPI, dysphagia or dysarthria
* Incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OSA patients who undergo a maxillomandibular advancement
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Nasality | Timpoints: T0 preoperative, T1 6 weeks after surgery, T2 3 months after surgery, T3 6 months after surgery, T4 1 year after surgery
  Nasality is measured using the Nasometer. The outcome consists of three scores: oral, nasal, and mixed. The nasality score is expressed as a percentage (0-100%), where a higher score indicates greater nasality. These scores will be compared across five time points.

SECONDARY OUTCOMES:
Swallowing | T0 preoperative, T1 6 weeks after surgery, T2 3 months after surgery, T3 6 months after surgery, T4 1 year after surgery
  FOIS (functional oral intake scale), swallow volume and swallow time will be evaluated by the speech therapist.
  The FOIS is used to describe the level of oral food and liquid intake in individuals with swallowing difficulties. The scale ranges from 0 to 7, where:
  0: Nothing by mouth (NPO) - the individual does not take any food or liquid orally.
  1. Tube dependent with minimal attempts of food or liquid - primarily tube-fed but may have some minimal oral intake.
  2. Tube dependent with consistent oral intake of food or liquid - mostly tube-fed but regularly takes some oral intake.
  3. Tube dependent with oral intake of food or liquid without special preparation - mostly tube-fed but oral intake is not modified.
  4. Total oral diet of a single consistency - the individual eats only one consistency of food or liquid.
  5. Total oral diet with multiple consistencies but requiring special preparation or compensations - eats various consistencies but with mod
Speech | T0 preoperative, T1 6 weeks after surgery, T2 3 months after surgery, T3 6 months after surgery, T4 1 year after surgery
  The Cleft Audit Protocol for Speech - Adult (CAPS-A) is a standardized assessment tool designed to evaluate speech outcomes in individuals with cleft lip and/or palate. It focuses on identifying speech characteristics commonly affected by cleft conditions, such as resonance, nasal emission, articulation, and overall speech intelligibility.
  What CAPS-A measures:
  Resonance: The degree of nasal quality in the voice (e.g., hypernasality or hyponasality).
  Nasal Emission: The presence of air escaping through the nose during speech, which can affect clarity.
  Articulation: Accuracy and clarity of speech sounds, especially those that may be distorted due to structural or functional issues.
  Overall Intelligibility: How well the speech can be understood by listeners.
  Outcome measures:
  CAPS-A uses a 5-point scale to rate the severity of certain speech characteristics, such as resonance and nasal emission, ranging from no impairment to severe impairment.
  Additionally, the presence or absen
Subjective outcomes: The Functional Outcomes of Sleep Questionnaire (FOSQ) | T0 preoperative, T1 6 weeks after surgery, T2 3 months after surgery, T3 6 months after surgery, T4 1 year after surgery
  Functional Outcomes of Sleep Questionnaire (FOSQ)
  The Functional Outcomes of Sleep Questionnaire (FOSQ) is a patient-reported outcome measure designed to assess the impact of excessive daytime sleepiness on daily activities and quality of life. It evaluates how sleep disorders affect a person's ability to carry out routine tasks and engage in social and occupational activities.
  What it measures:
  The FOSQ covers multiple domains including general productivity, activity level, vigilance, social outcomes, and intimacy/sexual relationships.
  It reflects the functional limitations caused by sleepiness rather than just sleep symptoms alone.
  Outcome measures:
  The FOSQ produces a total score and subscale scores for each domain. Scores typically range from 0 to 4 or 5 per item, with higher scores indicating better functional status and less impact of sleepiness.
  The total score summarizes overall functional status related to sleepiness, with lower scores reflecting greater impairment.
Subjective outcome: Neuro Sensory Disturbance Questionnaire | T0 preoperative T1 +6 weeks post op T2 +3 months post op T3 +6 months post op T4 +12 months post op
  Neuro Sensory Disturbance Questionnaire
  The Neuro Sensory Disturbance Questionnaire is used to assess sensory symptoms related to neurological conditions, such as numbness, tingling, burning, or altered sensation. It helps to quantify the presence and severity of sensory disturbances that may affect daily functioning.
  What it measures:
  The questionnaire evaluates the type, frequency, and intensity of sensory symptoms.
  It may also include questions on the impact of these symptoms on daily activities and quality of life.
  Outcome measures:
  Scores are often based on ordinal scales (e.g., 3- or 5-point scales) rating severity or frequency of symptoms.
  The questionnaire may provide subscale scores for different sensory modalities (e.g., pain, numbness).
  A total score can be calculated to reflect overall neuro-sensory disturbance, with higher scores indicating more severe or frequent symptoms.

OTHER OUTCOMES:
Descriptive data | Pre operative data extraction
  AHI = apnea/hypoapnea index:
  Normal: AHI < 5 events/hour Mild sleep apnea: AHI 5-14 events/hour Moderate sleep apnea: AHI 15-29 events/hour Severe sleep apnea: AHI ≥ 30 events/hour Higher AHI values indicate more severe sleep-disordered breathing.
  Age: in years
  BMI:
  Underweight: BMI < 18.5 Normal weight: BMI 18.5-24.9 Overweight: BMI 25-29.9 Obesity: BMI ≥ 30
  Gender: male/female

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be shared with other researches: speech therapist and my supervisor.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 01-06-2025 - 01-06-2028
Access Criteria: The speech therapist will have access to all data as she is responsible for conducting the measurements. I will also have access to all data since I am responsible for analyzing it and monitoring the study. My supervisor will have access to the outcomes, which are anonymized.

REFERENCES:
- [Background] Kummer AW, Marshall JL, Wilson MM. Non-cleft causes of velopharyngeal dysfunction: implications for treatment. Int J Pediatr Otorhinolaryngol. 2015 Mar;79(3):286-95. doi: 10.1016/j.ijporl.2014.12.036. Epub 2015 Jan 5. PMID 25604261
- [Background] Li KK, Troell RJ, Riley RW, Powell NB, Koester U, Guilleminault C. Uvulopalatopharyngoplasty, maxillomandibular advancement, and the velopharynx. Laryngoscope. 2001 Jun;111(6):1075-8. doi: 10.1097/00005537-200106000-00027. PMID 11404624
- [Background] Kummer AW. Types and causes of velopharyngeal dysfunction. Semin Speech Lang. 2011 May;32(2):150-8. doi: 10.1055/s-0031-1277717. Epub 2011 Sep 26. PMID 21948641